CLINICAL TRIAL: NCT02604940
Title: Evaluation of a Single Intra-operative Dose of Dexmedetomidine on Post-operative Narcotic Requirements and Pain Scores in Bariatric Surgery Patients
Brief Title: Evaluation of Dexmedetomidine on Post-operative Narcotic Requirements and Pain Scores in Bariatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Pavithra Ellison, Assistant Professor, Department of anesthesiology, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1306055796
Record Dates: First submitted 2015-10-14; First posted 2015-11-16 (Estimated); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Pain
Keywords: Postoperative narcotic requirements; Dexmedetomidine; Bariatric Surgery
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexmedetomidine (Experimental): Experimental group will receive 1mcg/kg IV dexmedetomidine over 10 minutes intraoperatively at the beginning of surgical closure
  Interventions: Drug: Dexmedetomidine
- Normal Saline (Active Comparator): Control group will receive Normal saline over 15 minutes at the beginning of surgical closure
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — 1mcg/kg IV dexmedetomidine over 10 minutes from 60ml syringe in OR upon notification of surgical closure
  Other Names: Precedex
  Arms: dexmedetomidine
Drug: Normal Saline — 60ml Saline delivered over 10 minutes in OR upon notification of surgical closure.
  Arms: Normal Saline

SUMMARY:
The purpose of the study is to determine whether a single bolus dose of dexmedetomidine administered during bariatric surgery has any effect on the amount of narcotic pain medications required by an individual after surgery. Patients who undergo weight loss surgery will be randomized into two groups - group one -dexmedetomidine group and group two- control group. Both groups will receive a standard anesthetic. Control group will receive weight based dose of fentanyl (standard narcotic pain reliever), intravenous acetaminophen (non-narcotic pain reliever), and 60ml saline. Experimental group will receive weight based dose of fentanyl (standard narcotic pain reliever), intravenous acetaminophen (non-narcotic pain reliever), and dexmedetomidine (given as 1mcg/kg over 10 minutes Intravenous). The Patient will then awaken after surgery in post anesthetic recovery unit and be given a patient controlled analgesia (PCA) pump with hydromorphone (long acting narcotic pain reliever). The amount of hydromorphone used will be recorded by the PACU nurse to the electronic health record ( routine practice) in the two groups and compared for pain medicine requirements. Secondary endpoints will be Visual Analog Score (VAS) pain score, respiratory rate, heart rate, blood pressure oxygen saturation and respiratory rate. All will be recorded at 30,60,90,120 and 240 minutes in the electronic medical record in PACU and compared between the two groups . All the data - Intra operative and Post -operative - Post Anesthesia Care Unit ( PACU) data will be retrieved from the electronic Medical record (EMR). All intra-operative data is automatically computed into the patients EMR. All PACU data is routinely entered into the EMR by the PACU nurse including the PCA data.

DETAILED DESCRIPTION:
This study will evaluate the postoperative opioid sparing effects of dexmedetomidine given as single bolus dose intraoperatively. Dexmedetomidine is an agonist of α2-adrenergic receptors sedative medication used by intensive care units and anesthesiologists and is unique in its ability to provide sedation without causing respiratory depression. Recently, it has received attention for its potential for additive analgesia. The study population will be patients undergoing gastric bypass surgery. The study population of bariatric surgery patients was chosen due to high prevalence of sleep apnea and Pickwickian component that can be worsened with opioid analgesia in the postoperative period. The purpose of the study is to test whether the use of a single bolus dose dexmedetomidine in addition to standard dose pain regimen decreases postoperative narcotic requirements when compared to standard dose pain regimen alone. The secondary purpose is to study whether single bolus dose dexmedetomidine reduces respiratory rate, heart rate, systolic and mean blood pressure, patient PCA demand bolus requests and VAS pain scores in the postoperative period. The overall goal of the study is to establish evidence of dexmedetomidine's role in multimodal pain relief in the bariatric surgery population with the possibility of other patient subgroups to follow

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing open bariatric surgery at WVUH-ruby hospital. - They must be ASA class 1, 2 and 3.
* Consented individuals.
* They must be between the age of 18 to 55.

Exclusion Criteria:

* History of bradycardia or tachy-brady syndrome HR<45.
* 1st degree heart block or higher.
* Patient refusal.
* On pain medication for any reason for more than 24 hrs within 2 weeks of procedure.
* Allergy to medication.
* History of alcohol or drug abuse.
* History of Cardiac/ liver/ kidney disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavithra Ranganathan, Principal Investigator — West Virginia University
Locations (1):
- WVU Healthcare Ruby Memorial Hospital, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ranganathan P, Ritchie MK, Ellison MB, Petrone A, Heiraty P, Tabone LE. A randomized control trial using intraoperative dexmedetomidine during Roux-en-Y gastric bypass surgery to reduce postoperative pain and narcotic use. Surg Obes Relat Dis. 2019 Apr;15(4):588-594. doi: 10.1016/j.soard.2019.01.021. Epub 2019 Jan 31. PMID 30824336

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine | Normal Saline
Started | 26 | 20
Completed | 26 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Normal Saline | Total
Number analyzed (Participants) | 26 | 20 | 46
Age, Continuous [Mean (Full Range); unit: years] | 45.1 [21 to 65] | 43.2 [25 to 59] | 44.3 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 46.0 [34.7 to 57.0] | 45.63 [35.7 to 59.1] | 45.89 [34.7 to 59.1]

OUTCOME MEASURES:

1. Primary Outcome: Quantity of Narcotic Utilized by Patient for Pain in Milligrams at 240 Minutes
Description: Amount of narcotic delivered to patient by Patient Controlled Analgesia (PCA)Pump in milligrams at 240 minutes
Time Frame: At 240 minutes after arriving in Post Anesthesia care Unit
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Dexmedetomidine | Normal Saline
Number analyzed (Participants) | 26 | 20
mg | 2.66 (2.02) | 3.7 (2.3)

2. Secondary Outcome: Pain Score on a Scale of 1-10 (1=Least 10= Worst)
Description: Pain scores on a scale of 1-10 measured in the post anesthesia care unit at 240 minutes
Time Frame: At 240 minutes after arriving in Post Anesthesia care Unit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine | Normal Saline
Number analyzed (Participants) | 26 | 20
score on a scale | 3.6 (2.8) | 6.7 (3)

3. Secondary Outcome: Heart Rate - Per Minute
Description: Heart Rate as recorded in the Medical record at 240 Minutes
Time Frame: At 240 minutes after arriving in Post Anesthesia care Unit
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Dexmedetomidine | Normal Saline
Number analyzed (Participants) | 26 | 20
beats per minute | 70 (12) | 86 (14)

4. Secondary Outcome: Blood Pressure - Measured in mmHg
Description: Blood Pressure as recorded in the Medical record at 240 Minutes
Time Frame: At 240 minutes after arriving in Post Anesthesia care Unit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine | Normal Saline
Number analyzed (Participants) | 26 | 20
mmHg
  Systolic BP | 107 (17) | 148 (16)
  Diastolic BP | 56 (15) | 79 (13)

5. Secondary Outcome: Oxygen Saturation - Measured in Percentage
Description: Oxygen Saturation as recorded in the medical record at 240 minutes
Time Frame: At 240 minutes after arriving in Post Anesthesia care Unit
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Dexmedetomidine | Normal Saline
Number analyzed (Participants) | 26 | 20
percentage of oxygen saturation | 97 (2) | 99 (2)

6. Secondary Outcome: Respiratory Rate as Measured Per Minute
Description: Breaths per minute as recorded in the medical record at 240 minutes
Time Frame: At 240 minutes after arriving in Post Anesthesia care Unit
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Dexmedetomidine | Normal Saline
Number analyzed (Participants) | 26 | 20
Breaths per minute | 17 (4) | 17 (3)

ADVERSE EVENTS:
Time Frame: Collected over 4 hours during PACU recovery
Description: PACU Standard of Care procedures
Arm/Group | Dexmedetomidine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/20
Other Adverse Events (participants affected / at risk) | 0/26 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-04-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT02604940/Prot_SAP_000.pdf
  • Informed Consent Form (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT02604940/ICF_001.pdf